CLINICAL TRIAL: NCT05163314
Title: A Phase 3, Prospective, Open-Label, Multisite, Extension of Phase 3 Studies To Assess the Long-Term Safety and Tolerability of Soticlestat as Adjunctive Therapy in Subjects With Dravet Syndrome or Lennox-Gastaut Syndrome (ENDYMION 2)
Brief Title: A Study of Soticlestat as an Add-on Therapy in Children and Adults With Dravet Syndrome or Lennox-Gastaut Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to negative results from phase 3 SKYLINE and SKYWAY studies and unrelated to patient safety it has been determined that supplementary data from TAK-935-3003 study is no longer necessary. Therefore, Takeda has made a decision to close this study
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-935-3003; 2021-002482-17 (EudraCT Number); jRCT2051210182 (Registry Identifier: jRCT); 2022-502802-34-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Dravet Syndrome (DS); Lennox Gastaut Syndrome (LGS)
Keywords: Drug Therapy
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome | interventions — soticlestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Soticlestat (Experimental): Participants with DS and LGS will receive:Participants weighing <45kg:Soticlestat,mini-tablets,titrated from lower dose level(60mg to 140mg) to higher dose(100mg to 200mg) twice daily(BID),based on body weight,orally/via enteral feeding tubes including but not limited to nasogastric(NG)-tube,gastrostomy tube(G-tube),MIC-KEY button,upto 2 weeks in Titration Period. Will continue to receive dose they are on at end of Titration Period,for approximately 4 years in Maintenance Period.Dose will be tapered down to lower dose(not less than lowest dose level based on weight)every 3 days until study drug is discontinued(upto 1week) in Taper Period.Participants weighing ≥45kg/adults:Soticlestat mini-tablets/tablets with starting dose of 200mg BID followed by 300mg BID,up to 2 weeks in Titration Period.Will continue to receive 300mg BID for approximately 4 years in Maintenance Period.Dose will be tapered down upto 100mg every 3 days until study drug is discontinued(up to 1 week) in Taper Period.
  Interventions: Drug: Soticlestat

INTERVENTIONS:
Drug: Soticlestat — Soticlestat mini-tablets or tablets
  Other Names: TAK-935

SUMMARY:
The main aim of the study is to learn if soticlestat, when given as an add-on therapy, reduces the number of seizures in children and adults with Dravet Syndrome (DS) or Lennox-Gastaut Syndrome (LGS).

Participants will receive their standard anti-seizure therapy, plus tablets of soticlestat. There will be scheduled visits and follow-up phone calls throughout the study.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat (TAK-935). Soticlestat administered long-term in pediatric and adult participants who participated in an antecedent soticlestat Phase 3 clinical study will be assessed for additional safety and tolerability data along with efficacy analysis, as well as palatability and acceptability of soticlestat in the pediatric population.

The study will enroll approximately 400 participants.

All participants will receive soticlestat based on their weight in the 2-week Titration Period (for participants who roll over from an antecedent double-blind study). Following the Titration Period, participants will continue to receive the same dose in the Maintenance Period. At the end of maintenance period, the dose will be down-tapered (unless already at the lowest dose) and then stopped. Participants not tolerating minimum dose of 100 mg twice a day (BID) will be discontinued from the study.

This multi-center trial will be conducted worldwide. The overall time to participate in the study will be approximately 4 years, or until the study is stopped at the discretion of the sponsor, or the product is approved and launched. Participants who discontinue study drug treatment before the completion of the study, will continue to be followed per protocol and maintain a daily seizure diary until the final follow-up phone call.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have:

* Been previously enrolled in a phase 3 soticlestat clinical study.

Exclusion Criteria:

1. Unstable, clinically significant neurologic (other than the disease being studied), psychiatric, cardiovascular, ophthalmologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, hematopoietic, endocrine disease, malignancy including progressive tumors, or other abnormality that may impact the ability to participate in the study or that may potentially confound the study results. It is the responsibility of the investigator to assess the clinical significance; however, consultation with the medical monitor may be warranted.
2. Abnormal and clinically significant ECG abnormality at Visit 1 including QT interval with Fridericia correction method (QTcF) >450 milliseconds (ms) confirmed with a repeat ECG using manual measurement of QTcF.
3. Participant is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property. Participants who have positive answers on item numbers 4 or 5 on the CSSRS before dosing are excluded. This scale will only be administered to participants aged ≥6 years.

Ages: 2 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 352 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants With At Least One Treatment Emergent Adverse Event (TEAE) | Up to 4 years
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug.
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Up to 4 years
  C-SSRS systematically tracks suicidal ideation and behavior. The total score range is 0 (no ideation is present) to 5 (active suicidal ideation with specific plan and intent). The higher the score, the greater one's suicidal ideation.
Change from Baseline in Body Weight for All Age Groups | Up to 4 years
Change from Baseline in Height for All Age Groups | Up to 4 years
Absolute Value for Tanner Stage for Children 6 to 17 Years of Age During the Study | Up to 4 years
  Tanner assessment score is used to document the stage of development of puberty by assessing the secondary sexual characteristics, rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size).
Absolute Value for Insulin-like Growth Factor 1 (IGF-1) for Children 2 to 17 Years of Age During the Study | Up to 4 years

SECONDARY OUTCOMES:
Percent Change from Baseline in Total Seizure Frequency per 28 Days for DS and LGS Participants | Up to 4 years
  Seizure frequency per 28 days is defined as total number of seizures reported during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline is defined as (frequency of seizures per 28 days during Treatment Period - frequency of seizures per 28 days at Baseline) divided by the frequency of seizures per 28 days at Baseline multiplied by 100.
Percent Change from Baseline in Convulsive Seizure Frequency per 28 Days in DS Cohort | Up to 4 years
  Convulsive seizure frequency per 28 days is defined as total number of convulsive seizures reported during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline will be defined as (frequency of convulsive seizures per 28 days during Treatment Period - frequency of convulsive seizures per 28 days at Baseline) divided by the frequency of convulsive seizures per 28 days at Baseline multiplied by 100.
Percent Change from Baseline in Major Motor Drop (MMD) Seizure Frequency per 28 Days in LGS Cohort | Up to 4 years
  MMD seizure frequency per 28 days is defined as total number of MMD seizures reported during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline will be defined as (frequency of MMD seizures per 28 days during the Treatment Period - frequency of MMD seizures per 28 days at Baseline) divided by the frequency of MMD seizures per 28 days at Baseline multiplied by 100.
Clinical Global Impression of Improvement (CGI-I) Score | Up to 4 years
  The CGI-I Clinician is a 7-point Likert scale that the investigator uses to rate a participant's change (improvement) in overall seizure control, behavior, safety and tolerability, after the initiation of study drug relative to Baseline (before treatment with study drug). The participant will be rated as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). Higher score will indicate worse symptoms.
Caregiver Global Impression of Improvement (Care GI-I) Score | Up to 4 years
  The Care GI-I is a 7-point Likert scale that the caregiver uses to rate improvement in overall seizure control, behavior, safety and tolerability after the initiation of study drug relative to Baseline (before treatment with study drug). The participant will be rated as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). The parent/caregiver will complete the Care GI-I via interview. Higher score will indicate worse symptoms.
CGI-I Seizure Intensity and Duration Score | Up to 4 years
  The CGI-I seizure intensity and duration instrument is used by the parent/caregiver to rate improvement in intensity and duration of convulsive seizures (DS Cohort) or MMD seizures (LGS Cohort) from Baseline. The participant's symptoms will be rated on 7-point scale as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). Higher score will indicate worse symptoms.
CGI-I Nonseizure Symptoms Score | Up to 4 years
  The CGI-I nonseizure symptoms instrument is a series of single-item assessments that the investigator uses to rate improvement in the symptoms and impacts in select nonseizure domains since initiating the study drug. The participant will be rated on 7-point scale by the investigator as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). At Baseline, a symptoms form is completed by the clinician in collaboration with the primary caregiver to assess the participants status based on the presence of any nonseizure symptoms. Higher score will indicate worse symptoms.
Change in Quality of Life Inventory-Disability (QI-Disability) Score | Up to 4 years
  The QI-Disability tool is a parent/caregiver-reported questionnaire that evaluates quality of life in children with intellectual disabilities. It contains 32 items covering 6 domains of quality of life: physical health, positive emotions, negative emotions, social interaction, leisure and the outdoors, and independence. Scores are from a 5-point Likert scale and then are transformed to a scale of 0 to 100. Possible scores range from 0-100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (116):
- United States (26):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Center For Neurosciences, Tucson, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California Benioff Children's Hospital, San Francisco, California
  - Colorado Children's Hospital, Denver, Colorado
  - Pediatric Neurology PA, Winter Park, Florida
  - Clinical Integrative Research Center of Atlanta, Atlanta, Georgia
  - Sunrise Pediatric Neurology, Marietta, Georgia
  - University of Iowa Hospitals & Clinics - (CRS), Iowa City, Iowa
  - Midatlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Minnesota Epilepsy Group PA, Saint Paul, Minnesota
  - Institute of Neurology and Neurosurgery at Saint Barnabas, LLC, Livingston, New Jersey
  - Boston Children's Health Physicians (BCHP), New York, New York
  - Northwell Health Physician Partners - Neurology at Lenox Hill, New York, New York
  - NYU Comprehensive Epilepsy Center, New York, New York
  - University of Toledo, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - WellSpan Oncology Research, York, Pennsylvania
  - Medical University of South Carolina Children Hospital - PIN, Charleston, South Carolina
  - Cook Children's Medical Center - Jane and John Justin Neurosciences Center, Fort Worth, Texas
  - University of Utah - Primary Children's Hospital - PPDS, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - MultiCare Institute for Research & Innovation (Tacoma), Tacoma, Washington
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Childrens Hospital, Brisbane, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - Centre Neurologique William Lennox, Ottignies-Louvain-la-Neuve, Brabant Wallon
  - Hopital Universitaire des Enfants Reine Fabiola, Brussels, Brussels Capital
- Brazil (5):
  - Instituto de Neurologia de Curitiba (INC), Curitiba, Paraná
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
  - Universidade de Sao Paulo, São Paulo
- Canada (2):
  - Child and Family Research Institute, Vancouver, British Columbia
  - Hospital For Sick Children, Toronto, Ontario
- China (12):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Children's Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Guangzhou Medical Univeristy, Guangzhou, Guangdong
  - Guangzhou Women And Children's Medical Center, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Wuhan Childrens hospital, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
- France (5):
  - Hopitaux de La Timone, Marseille, Bouches-du-Rhone
  - CHRU Dijon Hopital General, Dijon, Cote-d'Or
  - Hopital Roger Salengro, Lille, Nord
  - Hopital Necker - Enfants Malades, Paris
  - Hopital Robert Debre, Paris
- Germany (4):
  - Alberta Childrens Hospital, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum der Johann-Wolfgang Goethe-Universitat, Frankfurt am Main, Hesse
  - Krankenhaus Mara gGmbH - Epilepsiezentrum Bethel, Bielefeld, North Rhine-Westphalia
  - Kleinwachau Sachsisches Epilepsiezentrum Radeberg Gemeinnutzige Gmbh, Radeberg, Saxony
- Greece (4):
  - Childrens' Hospital of Athens 'P. and A. Kyriakou', Athens, Attica
  - Attikon University General Hospital, Chaïdári, Attica
  - University General Hospital of Larissa, Larissa
  - Hippokration Hospital, Thessaloniki
- Hungary (4):
  - Pecsi Tudomanyegyetem, Pécs, Baranya
  - Szent Janos Korhaz es Eszak-Budai Egyesitett Korhazak, Budapest
  - Bethesda Gyermekkorhaz, Budapest
  - Orszagos Klinikai Idegtudomanyi Intezet, Budapest
- Italy (6):
  - Ospedale Bellaria, Rome, Lazio
  - IRCCS Ospedale Pediatrico Bambino Gesu - INCIPIT - PIN, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - ASST di Mantova - Azienda Ospedaliera Carlo Poma, Mantova, Lombardy
  - ASST di Pavia - Fondazione Istituto Neurologico Mondino IRCCS, Pavia, Lombardy
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
- Japan (13):
  - Aichi Medical University Hospital, Nagakute-Shi, Aiti
  - Fukuoka Children's Hospital, Fukuoka, Hukuoka
  - Kanagawa Prefectural Hospital Organization Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Kumamoto-Ezuko Medical Center for The Severely Disabled, Kumamoto, Kumamoto
  - National Hospital Organization Nagasaki Medical Center, Omura-Shi, Nagasaki
  - National Hospital Organization Nishi-Niigata Chuo National Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Yasuhara Childrens Clinic, Neyagawa, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita-Shi, Osaka
  - National Hospital Organization Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - Hokkaido University Hospital, Chuo-Ku, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira-Shi, Tokyo
- Childrens University Hospital, Riga, Latvia
- Hospital Civil Fray Antonio Alcalde, El Retiro, Jalisco, Mexico
- Netherlands (2):
  - Kempenhaeghe - PPDS, Heeze, North Brabant
  - Stichting Epilepsie Instellingen Nederland, Zwolle, Overijssel
- Poland (4):
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - Dzieciecy Szpital Kliniczny im. Jozefa Polikarpa Brudzinskiego w Warszawie, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Kliniczny im. H.Swiecickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
- Russia (5):
  - Russian National Research Medical University n.a. N.I.Pirogov, Moscow, Moscow
  - Krasnoyarsk State Medical University n.a. V.F. Voyno-Ysenetskiy, Krasnoyarsk
  - Russian National Research Medical University n.a. N.I.Pirogov, Moscow
  - Tyumen State Medical Academy, Tyumen
  - UGMK-Zdorojie, LLC, Yekaterinburg
- Serbia (4):
  - Clinic for Neurology and Psychiatry for Children and Youth, Belgrade
  - Mother and Child Health Care Institute of Serbia Dr Vukan Cupic, Belgrade
  - University Clinical Center Nis, Niš
  - Children and Youth Health Care Institute of Vojvodina, Novi Sad
- Spain (6):
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Regional Universitario de Malaga Hospital General, Almería
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Vithas La Salud, Granada
  - Centro de Neurologia Avanzada, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Ukraine (5):
  - Municipal Institution Dnipropetrovsk Regional Children Clinical Hospital of DRC, Dnipro, Dnipropetrovsk Oblast
  - Communal Non-profit Enterprise Dnipro City Children Clinical Hospital #5 of DCC, Dnipro, Dnipropetrovsk Oblast
  - Communal Non-commercial Enterprise Iv-Frank Regional Childrens Clinical Hosp of Iv-Frank RC, Ivano-Frankivsk
  - CNPE Clinical Hospital Psychiatry of the Executive Body of the Kyiv City Council KCSA, Kyiv
  - SI Ukr. Med. Rehabilitation Center For Children With Organic Injury of Nervous System of MoH of Ukr, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/f1ef0bf231f449b6?idFilter=%5B%22TAK-935-3003%22%5D